CLINICAL TRIAL: NCT01639664
Title: COMPACT (COMbining Plasma-filtration and Adsorption Clinical Trial): Efficacy and Safety of High Doses CPFA (Coupled Plasma Filtration Adsorption) for Septic Shock in the ICU
Brief Title: COMPACT 2 - COMbining Plasma-filtration and Adsorption Clinical Trial 2
Acronym: COMPACT-2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The interim analysis requested by the EDSMC shows higher mortality for the CPFA group compared to the controls, particularly in the first days of treatment.
Sponsor: Gruppo Italiano per la Valutazione degli Interventi in Terapia Intensiva (Other)
Collaborators: Bellco Srl Mirandola, Italy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6233
Record Dates: First submitted 2012-07-06; First posted 2012-07-13 (Estimated); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2017-03

CONDITIONS: Shock, Septic
Keywords: septic shock; intensive care medicine; coupled plasma filtration-adsorption
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High doses CPFA (Experimental): High doses CPFA (coupled plasma-filtration adsorption) with AMPLYA™ (BELLCO ITALY): >0.20 L/kg/day of plasma treated in the first 3 days after randomization.
  Interventions: Device: High doses CPFA
- Control group (No Intervention): standard practice

INTERVENTIONS:
Device: High doses CPFA — High doses CPFA (coupled plasma-filtration adsorption) with AMPLYA™ (BELLCO ITALY): >0.20 L/kg/day of plasma treated in the first 3 days after randomization.
  Arms: High doses CPFA

SUMMARY:
The study objective is to clarify whether the application of high doses CPFA (coupled plasma-filtration adsorption) in addition to the current clinical practice is able to reduce hospital mortality in septic shock patients in intensive care unit (ICU).

DETAILED DESCRIPTION:
Septic shock is a life-threatening clinical condition characterized by cardiovascular failure as a consequence of infection. Septic shock frequently causes multi-organ failure in the ICU. For this reason the extracorporeal therapies for the treatment of renal failure have become widespread in the ICU and, at the same time, new extracorporeal depurative techniques have been developed for the removal of inflammatory mediators. One of these techniques is CPFA (coupled plasma-filtration adsorption) that uses a sorbent once the separation between plasma and blood has been obtained with a plasma filter. The study objective is to clarify whether the application of high doses CPFA in addition to the current clinical practice is able to reduce hospital mortality in septic shock patients in intensive care unit. Secondary objectives are the resolution of septic shock and the reduction of ICU LOS (length of stay).

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the ICU in septic shock
* All patients that develop septic shock while in the ICU

Exclusion Criteria:

* Age less than 14 years
* Pregnancy
* Estimated life expectancy (due to comorbidities) less than 90 days
* Presence of relative or absolute contraindications to CPFA
* Admission from an other ICU where the patient remained for more than 24 hours
* Absence of informed consent

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2013-09; Primary Completion 2017-10-23 (Actual); Study Completion 2017-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Livigni, MD, Principal Investigator — Ospedale San Giovanni Bosco, Torino, ITALY
Locations (13):
- Italy (13):
  - Ospedale Madonna delle Grazie, U.O. di Anestesia e Rianimazione, Matera, Basilicate
  - Ospedale Maurizio Bufalini, UO Anestesia Terapia Intensiva, Cesena, Emilia-Romagna
  - Ospedale Morgagni-Pierantoni, U.O. Anestesia e Rianimazione, Forlì, Emilia-Romagna
  - Ospedale A. Manzoni, U.O. Anestesia e Rianimazione 1, Lecco, Lombardy
  - Ospedale SS. Antonio e Biagio e C. Arrigo, Servizio Anestesia, Rianimazione e Terapia Antalgica, Alessandria, Piedmont
  - Ospedale Maggiore, Chieri, Piedmont
  - Ospedale Santa Croce, Moncalieri, Piedmont
  - CTO Maria Adelaide, I Servizio Anestesia e Rianimazione, Turin, Piedmont
  - Ospedale San Giovanni Bosco, Servizio Anestesia e Rianimazione B-DEA, Turin, Piedmont
  - AOU Careggi, Florence, Tuscany
  - Ospedali Riuniti Valdichiana Senese, U.O. di Anestesia e Rianimazione, Montepulciano, Tuscany
  - Ospedale SS. Cosma e Damiano, Servizio Anestesia e Rianimazione, Pescia, Tuscany
  - Ospedale Alta Val d'Elsa, Terapia Intensiva, Poggibonsi, Tuscany

REFERENCES:
- [Derived] Garbero E, Livigni S, Ferrari F, Finazzi S, Langer M, Malacarne P, Meca MCC, Mosca S, Olivieri C, Pozzato M, Rossi C, Tavola M, Terzitta M, Viaggi B, Bertolini G; GiViTI. High dose coupled plasma filtration and adsorption in septic shock patients. Results of the COMPACT-2: a multicentre, adaptive, randomised clinical trial. Intensive Care Med. 2021 Nov;47(11):1303-1311. doi: 10.1007/s00134-021-06501-3. Epub 2021 Oct 3. PMID 34601619
- [Derived] Milla P, Viterbo ML, Mosca S, Arpicco S. Chemical and microbiological stability, anticoagulant efficacy and toxicity of 35 and 90 mM trisodium citrate solutions stored in plastic syringes. Eur J Hosp Pharm. 2018 Oct;25(e2):e83-e87. doi: 10.1136/ejhpharm-2016-001094. Epub 2017 Jan 13. PMID 31157074
- See also: GiViTI web site — http://www.giviti.marionegri.it

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The interim analysis requested by the EDSMC shows higher mortality for the CPFA group compared to the controls, particularly in the first days of treatment. This result raise concern that the use of CPFA may cause harm or worsen the clinical condition of septic shock patients. For this reason we did not conclude the participant enrollment of the study.
  The COMPACT-2 study has been prematurely terminated as from 23/10/2017.
Groups:
- High Doses CPFA: High doses CPFA (coupled plasma-filtration adsorption) with AMPLYA™ (BELLCO ITALY): >0.20 L/kg/day of plasma treated in the first 3 days after randomization and on each of the subsequent days in which the patient is still in septic-shock condition.
Period: Overall Study
Arm/Group | High Doses CPFA | Control Group
Started | 63 | 52
Completed | 63 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Doses CPFA | Control Group | Total
Number analyzed (Participants) | 63 | 52 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 20 | 44
  >=65 years | 39 | 32 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (13.8) | 67.0 (10.5) | 67.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 40 | 28 | 68
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 63 | 52 | 115
Length of stay before ICU admission [Mean (Standard Deviation); unit: days] | 4.0 (7.2) | 3.0 (5.2) | 3.6 (6.4)
SAPS II [Median (Inter-Quartile Range); unit: units on a scale] — The Simplified Acute Physiology Score (SAPS II) is a severity score and mortality estimation tool developed from a large sample of medical and surgical patients in North America and Europe. SAPS II consists of 17 variables: 12 physiological variables, age, type of admission, and 3 variables related to underlying disease. For the physiological variables, the worst value during the first 24 hours of ICU admission is used for the calculation. The SAPS II results in a point score between 0 and 163 and a predicted mortality between 0% and 100%. Lower values are associated with lower mortality.
  units on a scale | 60 [45 to 73.8] | 55 [47.8 to 67.5] | 57.5 [46.75 to 72]
Septic shock on admission [Count of Participants; unit: Participants] | 45 | 40 | 85

OUTCOME MEASURES:

1. Primary Outcome: Hospital Mortality
Description: For patients discharged to other hospital, it will be intended as mortality at the discharge from the latest hospital in which the patients stayed.
Time Frame: At the discharge from the latest hospital (on average 30.3 days)
Measure: Count of Participants; unit: Participants
Groups:
- Control: Standard practice
Arm/Group | High Doses CPFA | Control
Number analyzed (Participants) | 63 | 52
Participants | 35 | 24

2. Secondary Outcome: Mortality Within 90 Days From Randomization
Time Frame: 90 days from randomization
Population: 11 patients lost at the follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | High Doses CPFA | Control Group
Number analyzed (Participants) | 56 | 48
Participants | 36 | 25

3. Secondary Outcome: ICU LOS Reduction Measured as Days Not Spent in the ICU During the First 30 Days From Randomization
Time Frame: 30 days from randomization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | High Doses CPFA | Control
Number analyzed (Participants) | 63 | 52
days | 6.6 (9.7) | 9.3 (9.9)

4. Secondary Outcome: Septic Shock Resolution Measured as Number of Days Free of Vasoactive Drugs From Randomization
Time Frame: 15 days from randomization
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All patients showing a serious adverse event probably related to the experimental technique were monitored until the symptoms disappear, or the laboratory values return to normal, or until a reasonable explanation of the observed changes emerges, or until death. In the last case, the pathologist report should be provided, whenever possible. Patients were monitored up to 90 days. All adverse events were recorded on an ad hoc form.
Description: In the field of intensive care medicine, the incidence of critical events during the stay in the ICU is high by definition. For this reason, only unfavorable and unintended sign (including abnormal laboratory finding), symptom, or disease probably related to the experimental technique has been taken into account. Non-treatment-related Adverse Events were not monitored.
Arm/Group | High Doses CPFA | Control Group
All-Cause Mortality (participants affected / at risk) | 36/63 | 25/52
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/52
Other Adverse Events (participants affected / at risk) | 0/63 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-01-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT01639664/Prot_SAP_000.pdf